CLINICAL TRIAL: NCT03991793
Title: Granzyme A in Patients With E. Coli Bacteremic Urinary Tract Infections
Acronym: GABEC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Responsible Party: Principal Investigator, José Ramón Paño Pardo, Principal Investigator. Assistant Professor, Instituto de Investigación Sanitaria Aragón
Other Study IDs: PI19/070
Record Dates: First submitted 2019-06-13; First posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Bloodstream Infection; Sepsis; Pathogenesis; Escherichia Coli Bacteremia
Keywords: Granzyme A; Sepsis; Pathogenesis; Escherichia coli Bloodstream Infection; Immunopathology
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (serum) for GZM A levels and gzmA polymorphisms E. coli strains
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis: Severe sepsis or septic shock (2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definition Conference)
- Control: Absence of severe sepsis or septic shock (2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definition Conference)

SUMMARY:
Background: Survival in Granzyme A gene (gzmA) knocked-out mice was significantly longer than in wild-type mice in a murine peritonitis model (cecal ligation puncture).

Hypothesis: GZM A has a pathogenic role in sepsis in humans and gzmA polymorphisms can help to predict the risk of sepsis among patients with systemic infections (E. coli bacteremic urinary tract infections).

Objectives:

1. To assess the correlation between GZM A serum levels and systemic inflammatory response in a human model of infection/sepsis (E. coli bacteremic UTI)
2. To characterize gzmA polymorphisms among patients with E. coli bacteremic UTI
3. To determine GZM A serum kinetics among patients with E. coli bacteremic UTI
4. To characterize E. coli strains causing bacteremic UTI: antimicrobial phenotype and virulence factors ("virulome").

Methods:

* Design and setting: Prospective nested case-control study
* Study population: consecutive adult patients with bacteremic urinary tract infections (UTIs) caused by E. coli
* Exclusion criteria: Patients with conditions that significantly compromise immune status or patients exposed to urologic procedures
* Estimated sample size: 50 patients with a sepsis/ non sepsis 1:1 ratio. Septic and non septic patients will be matched on gender, age (+/- 10 years), comorbidity (Charlson score +/-1), time symptom onset to blood culture (+/- 24h)
* Measurements: GZM A serum levels will be determined on day 0, day 2-3, day 30. GZM A kinetics, gzmA polymorphisms (whole exome sequencing).Whole genome sequencing of E. coli isolates retrieved from blood cultures will be performed.
* Analysis: Association between GZM A levels and gzmA polymorphisms and sepsis will be analyzed adjusting for patient, infection and microorganism-related factors (multivariate analysis).

DETAILED DESCRIPTION:
1. Research hypothesis

The research team has explored the role of GZM A

1. Conceptual hypothesis:

   * Granzyme A is a pathogenic sepsis mediator.
   * Granzyme A gene polymorphisms determine the serum concentration of GZM A in patients with systemic infections.
   * Granzyme A gene polymorphisms determine the risk of sepsis among patients with systemic infections.
2. Operational hypothesis:

   * Among patients with bacteremic (E. coli) urinary tract infections (UTIs), GZM A levels are significantly higher in those patients who develop sepsis as compared with those who do not develop sepsis.
   * There are significant differences in the GZM A gene polymorphism profile of patients with bacteremic (E. coli) UTIs who develop sepsis as compared with those who do not develop sepsis.

     2. Aims and objectives
   * Aims

     1. To assess the pathogenic role of GZM A in sepsis in patients with bacteremic (E. coli) UTIs.
     2. To explore the capability of GZM A polymorphisms to anticipate the risk of developing sepsis in patients with bacteremic (E. coli) UTIs.
     3. To evaluate the potential usefulness of GZM A as a diagnostic biomarker of sepsis in patients with bacteremic (E. coli) UTIs.
     4. To characterize E. coli "virulome" among circulating uropathogenic strains.
   * Objectives

     1. To evaluate the correlation between serum levels of GZM A and systemic inflammatory response in patients with bacteremic (E. coli) UTIs.
     2. To characterize GZM A gene polymorphisms among patients with bacteremic (E. coli) UTIs
     3. To assess GZM A serum kinetics among patients with bacteremic (E. coli) UTIs
     4. To phenotypically and molecularly characterize E. coli strains causing bacteremic UTIs, including their virulence factors ("virulome").

     3. Expected outcomes.
   * Characterization of the pathogenic role of GZM A in sepsis in patients with systemic infections
   * Characterization of GZM A as a sepsis biomarker in a human model of infection-sepsis.
   * Phenotypical and molecular characterization of uropathogenic E. coli causing bloodstream infections.

     4. Methods

   4.1. Design and project scope

   - Prospective, exploratory nested case-control study to be conducted at one academic hospital (Hospital Clínico Universitario Lozano Blesa) affiliated with the Instituto de Investigación Sanitaria Aragón (IIS Aragón).

   4.2. Study period: June 2019 - December 2020.

   4.3. Patients and sample size

   Inclusion criteria (To meet all):
   * Age >= 18 years old.
   * E. coli bloodstream infection
   * Urinary source. Urinary source should be considered if (any) of the following:

     1. Urinary source is clinically suspected and both E. coli isolates (in blood and in urine culture) share the same phenotype (antibiogram).
     2. Urinary source/origin is clinically suspected, and the urine culture is negative, but the patient had received at least one dose of any systemic antibiotic with antimicrobial activity against the E. coli strain causing the BSI before blood cultures were obtained.
     3. Both isolates (in blood and in urine culture) share the same phenotype (antibiogram) and there is no alternative source.

   Exclusion criteria:
   1. Use of systemic antibiotics for >48h in the two months preeeding the episode.
   2. Immunocompromised hosts - Patients receiving systemic steroid use (>10 mg prednisone/day during 10 or more days in the previous 2 months).

      * Patients receiving biological therapy (previous 2 months).
      * Active solid or hematological cancer.
      * HIV +.
      * Neutropenia < 500 PMN/microl.
   3. Basal urinary tract abnormalities or locally modified vesical microbiome (any):

      - Ureteroileostomy, ureterosigmoidostomy, ureterostomy (Bricker) or nephrostomy.
      * Indwelling urinary catheter (in the last two months)
      * Urological surgery (in the last two months).
      * Intravesical chemotherapy (in the last two months).
      * Intravesical BCG instillation (in the last two months).

      Potential candidates will be detected daily by the microbiologists on the research team. Inclusion criteria will be verified in the multidisciplinary meeting that antimicrobial stewardship teams (AST) conduct on a daily basis at the participating hospital.

      Estimated size of the study population. Matching:

      - 50 patients with a sepsis/ non sepsis 1:1 ratio will be included.

      - Septic and non-septic patients will be matched on gender, age (+/- 10 years), comorbidity (Charlson score +/-1), time symptom onset to blood culture (+/- 24h)

      4.4. Definitions

      Cases (sepsis / septic shock):

      - Sepsis or shock septic are defined as life-threatening organ dysfunction caused by a dysregulated host response to infection according to the 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definition Conference.

      Controls:

      - Absence of sepsis or septic shock according to the 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definition Conference.

      4.5. Variables

      4.5.1. Patient-related variables:

      - Demographical: gender, age.
      * Comorbidity: Modified Charlson Index
      * Baseline serum creatinine.

      4.5.2. Infection-related variables.

      - Time from the onset of symptoms to the start of antimicrobial treatment.

      - Time from the onset of symptoms to the start of appropriate antimicrobial treatment.

      - Time form the onset of symptoms to the surgical therapy (if needed).
      * Clinical severity at time 0 (blood culture), and day 2- 3 and day 30: sepsis score.

      4.5.3. Inflammation, sepsis mediators and biomarkers. - The following biomarkers will be determined during patient enrollment: - White blood cell count and differential. - Platelet count. - Fibrinogen. - Prothrombin activity.

      - C reactive protein.
      * Procalcitonin.
      * GZM A.

      GZM A serum levels will be obtained in all patients during the enrollment visit, the 2-3 day and the 30 day visits (GZM A kinetics). GZM A levels will be determined by an ELISA commercial assay (Human Granzyme A ELISA development kit{HRP]; Mabtech).

      GzmA gene polymorphisms, as well as other potentially associated mutations, will be screened by Whole Exome Sequencing (WES). To this aim, we will use DNA isolated from peripheral blood cells and the AmpliSeq technology kit on the Ion Torrent platform following the manufacturer's instructions. This platform is available at the Genomics Central Research Unit (CRU) at CIBA from University of Zaragoza/IIS Aragon. All kits for isolating and analyzing DNA samples are commercially available and optimized by Thermo Scientific. Bioninformatic analysis will be performed by an agreement established between Genomics CRU and Micromics SL led by Pedro Gonzalez at CRG in Barcelona.

      4.5.4. Microbiological variables
      * Minimum inhibitory concentrations (MIC) of the E. coli isolates retrieved from urine and blood cultures will be determined through automated microdilution panels as routinely performed by the Microbiology Laboratory of participating hospitals.
      * Whole genome sequencing (WGS) of the E. coli strains isolated in blood and urine cultures. The presence of E. coli known virulence factors will be analyzed and a virulence score for each strain will be calculated (Mora-Rillo et al., 2015).

ELIGIBILITY:
Inclusion Criteria:

* E. coli bacteremic urinary tract infection

Exclusion Criteria:

* Immunocompromised hosts: HIV/AIDS, Neutropenia, Solid neoplasia, Hematological neoplasia, patients receiving immunosuppressive therapy
* Systemic antibiotic therapy in the 2 months preceding the bloodstream infection
* Anatomical or functional urological abnormalities that require urological procedures in the previous 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with E. coli bloodstream infection from a urinary source
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-06-20 (Estimated); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Granzyme A serum levels | day 0
  GZM A serum concentration (GZM A serum levels) will be determined at day 0 by an ELISA commercial assay (Human Granzyme A ELISA development kit; Mabtech)

SECONDARY OUTCOMES:
gzmA polymorphisms | day 0
  GzmA gene polymorphisms, as well as other potentially associated mutations, will be screened by Whole Exome Sequencing (WES). To this aim, we will use DNA isolated from peripheral blood cells and the AmpliSeq technology kit on the Ion Torrent platform following the manufacturer's instructions. This platform is available at the Genomics Central Research Unit (CRU) at CIBA from University of Zaragoza/IIS Aragon. All kits for isolating and analyzing DNA samples are commercially available and optimized by Thermo Scientific.
Granzyme A serum kinetics | day 2-3 and day 30
  Granzyme A serum concentration will be determined at three time points: day 0, day 2-3 and day 30. GZM A serum concentration (GZM A serum levels) will be determined by an ELISA commercial assay (Human Granzyme A ELISA development kit; Mabtech)

CONTACTS AND LOCATIONS:
Overall Officials: José Ramón P Paño-Pardo, Principal Investigator — Instituto de Investigación Sanitaria Aragon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Arias MA, Jimenez de Bagues MP, Aguilo N, Menao S, Hervas-Stubbs S, de Martino A, Alcaraz A, Simon MM, Froelich CJ, Pardo J. Elucidating sources and roles of granzymes A and B during bacterial infection and sepsis. Cell Rep. 2014 Jul 24;8(2):420-9. doi: 10.1016/j.celrep.2014.06.012. Epub 2014 Jul 10. PMID 25017060
- [Result] Garcia-Laorden MI, Stroo I, Terpstra S, Florquin S, Medema JP, van T Veer C, de Vos AF, van der Poll T. Expression and Function of Granzymes A and B in Escherichia coli Peritonitis and Sepsis. Mediators Inflamm. 2017;2017:4137563. doi: 10.1155/2017/4137563. Epub 2017 Jun 12. PMID 28694562

DOCUMENTS (1):
  • Study Protocol (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT03991793/Prot_000.pdf